CLINICAL TRIAL: NCT01504685
Title: Long-Term Results of a Randomized Trial Comparing Banded-versus-Standard Laparoscopic Roux-en-Y Gastric Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Miguel F Herrera, Miguel F. Herrera, M.D., Ph.D., Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: banded/unbandedBypassINNSZ
Record Dates: First submitted 2012-01-02; First posted 2012-01-05 (Estimated); Last update posted 2012-01-26 (Estimated); Status verified 2012-01

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Obesity surgery; Gastric bypass; Banded gastric bypass
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unbanded laparoscopic gastric bypass (Active Comparator): Laparoscopic Roux- en-Y gastric bypass without any band around de gastric reservoir
  Interventions: Procedure: Unbanded Laparoscopic Roux- en-Y gastric bypass
- Banded laparoscopic gastric bypass (Active Comparator): Placement of a premeasured band or ring around the gastric reservoir, adjacent to the gastroenterostomy.
  Interventions: Procedure: Banded Laparoscopic Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Banded Laparoscopic Roux-en-Y gastric bypass — A 6.5-cm polypropylene Marlex mesh was placed immediately cephalad to the gastrojejunostomy. The gastrojejunostomy was hand-sewn in 2 layers using 3-0 Polyglactin for the internal and 3-0 silk for the external layer.
  The length of alimentary and biliopancreatic limbs was approximately 150 cm and 50 cm, respectively.
  Other Names: BLRYGB; banded gastric bypass
  Arms: Banded laparoscopic gastric bypass
Procedure: Unbanded Laparoscopic Roux- en-Y gastric bypass — A hand-sewn gastrojejunostomy in 2 layers using 3-0 Polyglactin for the internal and 3-0 silk for the external layer.
  To ensure a diameter of 1-1.5 cm,a 32F bougie was used to calibrate the gastro jejunum anastomosis. The length of alimentary and biliopancreatic limbs was approximately 150 cm and 50 cm, respectively.
  Other Names: Gastric bypass; LRYGB
  Arms: Unbanded laparoscopic gastric bypass

SUMMARY:
The purpose of the study is comparatively analyze the advantages and disadvantages of banded versus unbanded laparoscopic Roux-en-Y gastric bypass (RYGB).

The outcome variables of the general study included morbidity, maximal weight loss, and late weight regain.

DETAILED DESCRIPTION:
Obesity is a public health problem that has grown exponentially worldwide. Bariatric surgery has been recognized as the most effective treatment for morbid obesity. However, the debate about the best surgical procedure is still considerable.

Among a wide range of operations that have been used for morbid obesity, Roux-en-Y gastric bypass (RYGB) has shown an appropriate risk/benefit balance and has achieved a high degree of acceptance in America.

The weight loss pattern in RYGB is characteristic and includes significant eight loss during the first 2 years after surgery, followed by some weight regain after the second or third postoperative year. To prevent this some authors suggest the placement of a premeasured band or ring around the gastric reservoir, adjacent to the gastroenterostomy. This procedure has been called banded RYGB.

ELIGIBILITY:
Inclusion Criteria:

* body mass index of 40-55 kg/m2
* agreed to participate in this study with informed consent signed

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-05; Primary Completion 2005-03 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative morbidity | up to 5 years
  determine any morbidity related to the surgical procedure through the 5 years follow up
Change from Baseline weight assessed at different time points to determine maximal weight loss, | 3,6,9 months and 1,2,5 years
  determine changes in weight loss through 5 years follow up, measuring maximal weight loss.
Changes in weight assessed at different time points to determine weight regain | 3,6,9 months and 1,2,5 years
  identify changes in weight regain during the postoperative 5 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Miguel F Herrera, MD., PhD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutrición "Salavador Zubirán"